CLINICAL TRIAL: NCT02817321
Title: Thoracic Paravertebral Block : Effect on Acute Pain and Chronic Pain of Hepatectomy With Right J-shape Subcostal Incision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cui Xulei (Other)
Responsible Party: Sponsor-Investigator, Cui Xulei, Attending physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: cuixulei2
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Hepatectomy; Analgesia; Nerve Block
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine; isopropyl cyanoacrylate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-injection TPVB +continuous TPVB (Experimental): Single-injection of TPVB is given preoperatively followed with continuous infusion+ postoperative IPCA.
  Interventions: Procedure: single-injection TPVB + continuous TPVB; Device: Philip CX50 Ultrasound Scanner; Device: PAJUNK Contiplex S Catheter; Drug: single dose ropivacaine; Drug: continuously infusion of ropivacaine; Drug: Morphine given as IPCA
- IPCA (Active Comparator): postoperative IPCA is given alone
  Interventions: Drug: Morphine given as IPCA

INTERVENTIONS:
Procedure: single-injection TPVB + continuous TPVB — Inject local anesthetics in the T8 paravertebral space followed with catheter insertion and continuous local infusion.
  Arms: Single-injection TPVB +continuous TPVB
Device: Philip CX50 Ultrasound Scanner — The curved (C1-5) probe of Philip CX 50 Ultrasound Scanner is used for scanning
  Arms: Single-injection TPVB +continuous TPVB
Device: PAJUNK Contiplex S Catheter
  Arms: Single-injection TPVB +continuous TPVB
Drug: single dose ropivacaine — * 2mg/kg ropivacaine in saline with 1:200,000 adrenaline, 25ml in total
  * given immediately after the correct position of the tip of the needle has been confirmed
  Arms: Single-injection TPVB +continuous TPVB
Drug: continuously infusion of ropivacaine — * 0.2% ropivacaine, pulse dosadge: 0.125ml/kg/pulse, 1pulse/h at a rate of 6ml/minutes
  * given through the catheter inserted in the T8 paravertebral space following the single dose
  Arms: Single-injection TPVB +continuous TPVB
Drug: Morphine given as IPCA — bolus: 2mg, lock time: 10min, 1h limitation: 8mg

SUMMARY:
This prospective, randomized study,control study aims to compare the analgesic effect,opioids consumption,quality of recovery,length of hospital stay and incidence of chronic pain,et al. single-injection TPVB +continuous(pulsatile infusion) TPVB and intravenous patient-controlled analgesia (IPCA) alone in patients undergoing hepatectomy with right J-shape subcostal incision.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo hepatectomy with J-shape subcostal incision
* Informed consent

Exclusion Criteria:

* A known allergy to the drugs being used
* Coagulopathy, on anticoagulants
* Analgesics intake, history of substance abuse
* Participating in the investigation of another experimental agent
* Inability to properly describe postoperative pain to investigators (eg, language barrier, neuropsychiatric disorder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
cumulative morphine consumption | within 48 postoperative hours

SECONDARY OUTCOMES:
The pain scores determined by the numeric rating scale (NRS, 0-10) | At 0, 2,4, 8, 12, 24 ,48,72hours and 7day after the surgery
nausea and vomiting score | At 0, 2,4, 8, 12, 24 and 48hours after the surgery
pruritus score | At 0, 2,4, 8, 12, 24 and 48hours after the surgery
ambulation time | within the 7 days after surgery
time of recovery of bowl movement | within the 7 days after surgery
Postoperative hospital length of stay | Up to 4 weeks
patient satisfaction with anesthesia | 48 hours after surgery
  use the Chinese version Bauer questionnaire to assess the patient satisfaction with anesthesia
data collection of chronic pain | at 3,6,12 months after surgery
  Patients undergo a telephone interview with a questionnaire at 3, 6 and 12 months after surgery, the incidence and severity of chronic pain is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, MD., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Xulei CUI, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No